CLINICAL TRIAL: NCT04826016
Title: A Phase Ib/II Study to Optimize POL6326 (Balixafortide) in Combination With Nab-paclitaxel or Eribulin in Patients With HER2-negative Advanced Breast Cancer
Brief Title: POL6326 (Balixafortide) Plus Nab-paclitaxel or Eribulin in Patients With HER2-negative Advanced Breast Cancer
Acronym: POLTER
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funder decision
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP238; 2020-004203-13 (EudraCT Number)
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — balixafortide; eribulin; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PHASE Ib - ARM A: POL6326 (balixafortide) + eribulin (Experimental): On day 1 and 8 of each 21-day cycle (+/- 1 day) fixed eribulin dose of 1.23 mg/m2 (equivalent to 1.4 mg/m2 eribulin mesylate) combined with increasing doses of POL6326 (balixafortide) starting at a dose of 11 mg/Kg will be administered both intravenously. POL6326 (balixafortide) will be administered following a biphasic regimen (0,5 mg/Kg of POL6326 (balixafortide) dose during the first 30 min of treatment, the remaining dose during the following 3 h and 30 min for a total of 4h. Eribulin will be administered within 45 min after the end of the POL6326 (balixafortide) infusion over 2 to 5 min. Up to 4 additional cohorts may be introduced
  Interventions: Drug: POL6326; Drug: Eribulin
- PHASE Ib - ARM B: POL6326 (balixafortide) + nab-paclitaxel (Experimental): On day 1, 8 and 15 of each 28-day cycle (+/- 1 day) fixed nab-paclitaxel dose of 100 mg/m2 combined with increasing doses of POL6326 (balixafortide) starting at a dose of 5.5 mg/Kg will be administered both intravenously. POL6326 (balixafortide) will be administered following a biphasic regimen (0,5 mg/Kg of POL6326 (balixafortide) dose during the first 30 min of treatment, the remaining dose during the following 3 h and 30 min for a total of 4h. Nab-paclitaxel will be administered within 45 min after the end of the POL6326 (balixafortide) infusion over 30 min. Up to 5 additional cohorts may be introduced
  Interventions: Drug: POL6326; Drug: Nab paclitaxel
- PHASE 2 - ARM A: POL6326 (balixafortide) + eribulin (Experimental): MTD/RDP2 POL6326 (balixafortide) (from arm A phase Ib) will be administered over 4h intravenous infusion (biphasic regimen as detailed above/ phase Ib) followed by 1.4 mg/m2 eribulin over 5 min Intravenous infusion on days 1 and 8 in 21-day cycles (+/- 1 day).
  Interventions: Drug: POL6326; Drug: Eribulin
- PHASE 2 - ARM B: POL6326 (balixafortide) + nab-paclitaxel (Experimental): MTD/RDP2 POL6326 (balixafortide) (from arm B phase Ib) will be administered over 4h intravenous infusion (biphasic regimen as detailed above/ phase Ib) followed by 100 mg/m2 nab-paclitaxel over 30 min Intravenous infusion on days 1, 8 and 15 in 28-day cycles (+/- 1 day).
  Interventions: Drug: POL6326; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: POL6326 — POL6326 (balixafortide): starting dose at 5.5 mg/Kg. Intravenous administration on day 1 and 8 of each 21-day cycle (+/- 1 day) (Phase Ib ARM A and Phase II ARM A ) or on day 1, 8 and 15 of each 28-day cycle (Phase Ib ARM B and Phase 2 ARM B) (+/- 1 day).
  Other Names: Balixafortide
Drug: Eribulin — Eribulin: 1.23 mg/m2 (equivalent to 1.4 mg/m2 eribulin mesylate). Intravenous administration on day 1 and 8 of each 21-day cycle (+/- 1 day) (Phase Ib ARM A and Phase II ARM A ) or on day 1, 8 and 15 of each 28-day cycle (Phase Ib ARM B and Phase 2 ARM B) (+/- 1 day).
  Other Names: Halaven
  Arms: PHASE 2 - ARM A: POL6326 (balixafortide) + eribulin; PHASE Ib - ARM A: POL6326 (balixafortide) + eribulin
Drug: Nab paclitaxel — Nab-paclitaxel: 100 mg/m2. Intravenous administration on day 1 and 8 of each 21-day cycle (+/- 1 day) (Phase Ib ARM A and Phase II ARM A) or on day 1, 8 and 15 of each 28-day cycle (Phase Ib ARM B and Phase 2 ARM B) (+/- 1 day).
  Other Names: Abraxane
  Arms: PHASE 2 - ARM B: POL6326 (balixafortide) + nab-paclitaxel; PHASE Ib - ARM B: POL6326 (balixafortide) + nab-paclitaxel

SUMMARY:
This is a multicenter Phase Ib/II, open-label, dose-escalation study to optimize POL6326 (balixafortide) in combination with nab-paclitaxel or eribulin in patients with HER2-negative advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients ≥18 years of age with histologically confirmed invasive breast cancer.
2. Able to understand and willing to sign an IRB/IEC approved written informed consent document.
3. Locally advanced stages IIIB/C or metastatic stage IV disease by American Joint Committee on Cancer (AJCC) criteria (8th edition).
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Life expectancy greater than 12 weeks.
6. At least one measurable lesion per RECIST v.1.1 criteria.
7. Documented HER2-negative breast cancer in the advanced setting, with any ER and PgR status. HER2-negative (immunohistochemistry (IHC) 0, 1 or IHC 2+ and negative by in situ hybridization (ISH) test) status based on local testing on the most recent analyzed biopsy.
8. Prior Therapies:

   For POL6326 (balixafortide)-eribulin combination
   * phase Ib: At least 1 but no more than 3 prior chemotherapy-based lines of treatment for advanced or metastatic disease.
   * phase 2: At least 1 but no more than 2 prior chemotherapy-based lines of treatment for advanced or metastatic disease.

   Prior therapy should have included an anthracycline and a taxane, unless contraindicated based on investigator's criteria. Chemotherapy line given as (neo)adjuvant treatment will be considered a prior line of therapy if disease progression occurred within 12-months after completion of prior (neo)adjuvant therapy.

   Note: for phase Ib and phase 2: Disease progression after last systemic therapy documented by computerized tomography (CT) scan or magnetic resonance imaging (MRI). Exclusive tumor marker elevation will not be considered sufficient for diagnosis of disease progression.

   For POL6326 (balixafortide)-nab-paclitaxel combination
   * phase Ib: At least 1 but no more than 2 prior chemotherapy-based lines of treatment for advanced or metastatic disease.
   * phase 2: Up to 1 prior chemotherapy-based line of treatment for advanced or metastatic disease.

   For both combinations
   * phase Ib: patients with HR+ status (ER+ and/or PgR+) must have been treated with at least one line of endocrine therapy (or considered by the treating physician not to be a candidate for endocrine therapy).
   * phase 2: patients with HR+ status (ER+ and/or PgR+) must have been treated with at least one line of endocrine therapy and CDK4/6 inhibitors (unless contraindicated or not accessible).
9. At least 21 days from the completion of any previous cytotoxic chemotherapy or biological therapy at time of initiation of POL6326 (balixafortide).
10. Willingness and ability to provide a tumor biopsy from a newly obtained core or excisional biopsy not previously irradiated at the time of the inclusion and at the time of progression (optional) in order to perform exploratory studies. This enrolment criterium is optional for the dose-escalation part of the study, but mandatory for the final dose expansion (MTD/RP2D) cohorts. If this is not feasible (e.g., inaccessible tumor or subject safety concern), archival metastatic tumor samples might be acceptable after agreement with the Sponsor.
11. Willingness and ability to provide blood samples for exploratory studies as per study protocol.
12. Resolution of all acute toxic effects of prior anti-cancer therapy to grade 1 as determined by the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v. 5.0 criteria (except for alopecia or other toxicities not considered a safety risk for the patient at Investigator's discretion).
13. Adequate hematologic and organ function within 28 days before the first study treatment on Cycle 1 Day 1, defined by the following:

    * Hematological: White blood cell (WBC) count > 3.0 x 109/L, absolute neutrophil count (ANC) > 1.5 x 109/L phase Ib of the study, platelet count > 100.0 x109/L, and hemoglobin > 9.0 g/dL.
    * Hepatic: Serum albumin ≥ 3 g/dL; Total bilirubin ≤ 1.5 times the upper limit of normal (× ULN) (≤ 3 x ULN in the case of Gilbert's disease); aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 × ULN (in the case of liver metastases ≤ 5 × ULN); alkaline phosphatase (ALP) ≤ 3.0 × ULN (≤ 5 × ULN in the case of liver and/or bone metastases).
    * Renal: creatinine clearance ≥ 40 mL/min based on Cockcroft-Gault glomerular filtration rate estimation for POL6326 (balixafortide).
    * Coagulation: International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless on medication known to alter INR and/or aPTT.

For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive methods, or two effective contraceptive methods, as defined in the CSP during the treatment period and for at least 90 days after the last dose of study treatment, whichever is longer, and agreement to refrain from donating eggs during this same period. Women of childbearing potential must have a negative serum pregnancy test within 7 days before study treatment initiation

Exclusion criteria:

Patients will be excluded from the study if they meet ANY of the following criteria:

1. Eribulin-based combination: patients have previously received eribulin.
2. Peripheral neuropathy > Grade 1.
3. Prior radiotherapy to only site of disease.
4. Patients under concurrent local radiotherapy for pain control or life-threatening situations (e.g., spinal cord compression).
5. Known active uncontrolled or symptomatic CNS metastases as indicated by clinical symptoms, cerebral edema, and/or progressive growth. Patients with a history of CNS metastases are eligible if they have been definitively treated (e.g., radiotherapy, stereotactic surgery), and are clinically stable at least 4 weeks after completion of radiation therapy and/or surgery. Stable is defined as absence of new neurological symptoms, absence of need for dexamethasone or anticonvulsants, and radiographic confirmation of stable disease (SD). Radiographic confirmation of SD 4 weeks after completion of radiation therapy is not required unless indicated by neurological exam.
6. Presence of carcinomatous meningitis or leptomeningeal disease.
7. Therapeutic radiation therapy within 14 days (seven days for limited-field palliative radiotherapy) prior to study enrollment, or patients who have not recovered from radiotherapy-related toxicities to grade ≤ 1.
8. History of allergic reactions or known hypersensitivity attributed to compounds of similar chemical or biologic composition to POL6326 (balixafortide), eribulin or nab-paclitaxel, or to recombinant proteins, or any excipient contained in the drug formulation for POL6326 (balixafortide), eribulin or nab-paclitaxel.
9. Breastfeeding or pregnancy as determined by a serum pregnancy test (β-HCG) at screening, prior to the administration of POL6326 (balixafortide) and/or eribulin and/or nab-paclitaxel. Since β-HCG over expression can be also elevated in some tumor types, a positive result should be confirmed with a validated alternative test (e.g., ultrasound).

   Note: Postmenopausal women must have been amenorrhoeic for ≥ 12 months in order to be considered "of non-childbearing potential". This should be documented appropriately in the patient's medical history. More frequent assessments may be performed if medically indicated as determined by the study site Investigator, and these evaluations should be recorded in the CRF (Case Report Form).
10. Known HIV positivity on combination antiretroviral therapy.
11. Congenital long QT syndrome (LQTS) with corrected QT interval using the Fridericia formula (QTcF) ≥ 480 ms on baseline EKG.
12. Patients under treatment with drugs known to potentially prolong the QT interval, including class Ia and III anti-arrhythmic drugs will be either monitored for corrected QT (QTc) prolongation or excluded from participation in the trial, at the discretion of the treating physician.
13. Aany other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment contraindicate patient participation in the clinical study.
14. Severe concurrent psychiatric illness/social situation.
15. Concurrent malignancy or malignancy within five years of study enrollment with the exception of carcinoma in situ of the cervix, non-melanoma skin carcinoma, or stage I uterine cancer. For other cancers considered to have a low risk of recurrence, discussion with the Sponsor's Medical Monitor is required.
16. Treatment with approved or investigational cancer therapy within 21 days prior to initiation of study.
17. Concurrent participation in other clinical trial, except other translational studies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
PHASE Ib: Maximum tolerated dose (MTD) / Recommended phase II dose (RP2D) of POL6326 (balixafortide) | 12 - 24 months
  MTD/RP2D, based on the incidence of Dose limiting toxicities (DLT) defined as the highest dose level explored at which up to one third of evaluable patients develop a DLT during the first treatment cycle.
PHASE 2: Progression free survival (PFS) | from treatment initiation until objective tumor progression or death (at least 4.5 months)
  To assess the efficacy of POL6326 (balixafortide) in combination with either eribulin or nab-paclitaxel in terms of PFS as per RECIST v. 1.1 in patients with HER2-negative ABC.

SECONDARY OUTCOMES:
PHASE Ib: PFS | from treatment initiation until objective tumor progression or death (at least 4.5 months)
  To assess the efficacy of POL6326 (balixafortide) in combination with either eribulin or nab-paclitaxel in terms of PFS as per RECIST v. 1.1 in patients with HER2-negative ABC.
PHASE Ib: Overall response rate (ORR) | from baseline until end of study (will occur when all patients have discontinued treatment or 12 month after the last patient was enrolled on the study plus the safety follow up window of 28 days after last dose of study treatment in the last patient)
  To assess the preliminary efficacy of POL6326 (balixafortide) in combination with either eribulin or nab-paclitaxel in terms of ORR defined as the proportion of patients with complete response (CR) or partial response (PR) as per RECIST v.1.1
PHASE Ib: clinical benefit rate (CBR) | at least 6 months
  To assess the preliminary efficacy of POL6326 (balixafortide) in combination with either eribulin or nab-paclitaxel in terms of CBR, defined as the proportion of patients who obtain an objective response (CR or PR), or SD for at least 6 months for both combinations of the POL6326 (balixafortide) as per RECIST v.1.1.
PHASE IB: duration of response (DoR) | from the first occurrence of a documented objective response to disease progression or death, up to 12 months
  To assess the preliminary efficacy of POL6326 (balixafortide) in combination with either eribulin or nab-paclitaxel in terms of DoR, defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first, as per Investigator assessment using RECIST v.1.1.
PHASE Ib: maximum tumor shrinkage (MTS) | from baseline until end of study (will occur when all patients have discontinued treatment or 12 month after the last patient was enrolled on the study plus the safety follow up window of 28 days after last dose of study treatment in the last patient
  To assess the preliminary efficacy of POL6326 (balixafortide) in combination with either eribulin or nab-paclitaxel in terms of MTS, from baseline in the size of target tumor lesions, defined as the biggest decrease, or smallest increase if no decrease observed, as per RECIST v.1.1.
PHASE 2: ORR | from baseline until end of study (will occur when all patients have discontinued treatment or 12 month after the last patient was enrolled on the study plus the safety follow up window of 28 days after last dose of study treatment in the last patient)
  To assess the efficacy, of POL6326 (balixafortide) in combination with either eribulin or nab-paclitaxel in terms of ORR, defined as the proportion of patients with CR or PR, as per RECIST v.1.1.
PHASE 2: CBR | at least 6 months
  To assess the efficacy, of POL6326 (balixafortide) in combination with either eribulin or nab-paclitaxel in terms of CBR, defined as the proportion of patients who obtain an objective response (CR or PR), or stable disease for at least 6 months for both combinations of the POL6326 (balixafortide) as per RECIST v.1.1.
PHASE 2: time to response (TTR) | from treatment initiation to time of the first objective tumor response up to 12 months
  To assess the efficacy, of POL6326 (balixafortide) in combination with either eribulin or nab-paclitaxel in terms of TTR, defined as the time from treatment initiation to time of the first objective tumor response (tumor shrinkage of ≥ 30%) in patients who achieved a CR or PR, as per using RECIST v.1.1.
PHASE 2: DoR | from the first occurrence of a documented objective response to disease progression or death, up to 12 months
  To assess the efficacy, of POL6326 (balixafortide) in combination with either eribulin or nab-paclitaxel in terms of DoR, defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first, as per Investigator assessment using RECIST v.1.1.
PHASE 2: overall survival (OS) | from baseline until end of study (will occur when all patients have discontinued treatment or 12 month after the last patient was enrolled on the study plus the safety follow up window of 28 days after last dose of study treatment in the last patient
  To assess the efficacy, of POL6326 (balixafortide) in combination with either eribulin or nab-paclitaxel in terms of OS, defined as the time from treatment initiation to death from any cause.
PHASE 2: MTS | from baseline until end of study (will occur when all patients have discontinued treatment or 12 month after the last patient was enrolled on the study plus the safety follow up window of 28 days after last dose of study treatment in the last patient
  To assess the efficacy, of POL6326 (balixafortide) in combination with either eribulin or nab-paclitaxel in terms of MTS from baseline in the size of target tumor lesions, defined as the biggest decrease, or smallest increase if no decrease observed, as per RECIST v.1.1.
PHASE Ib/ PHASE 2: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of POL6326 (balixafortide) in combination with either eribulin or nab-paclitaxel | from baseline until end of study.All patients must be followed for AEs and SAEs for 28 days following the last dose of study drug
  Incidence and severity of AEs and SAEs according to the NCI-CTCAE v.5.0, including dose reductions, delays, and treatment discontinuations.
PHASE Ib - PHARMACOKINETICS (PK) in terms of area under the curve (AUC) | At the end of Cycle 1 (each cycle is 28 days in POL6326 (balixafortide) - eribulin combination and 21 days in POL6326 (balixafortide) - nab paclitaxel combination)
  Plasma PK parameter AUC of POL6326 (balixafortide)
PHASE Ib - PK in terms of clearance (CL), | At the end of Cycle 1 (each cycle is 28 days in POL6326 (balixafortide) - eribulin combination and 21 days in POL6326 (balixafortide) - nab paclitaxel combination)
  Plasma PK parameter CL of POL6326 (balixafortide)
PHASE Ib - PK in terms of distribution volume (Vd) | At the end of Cycle 1 (each cycle is 28 days in POL6326 (balixafortide) - eribulin combination and 21 days in POL6326 (balixafortide) - nab paclitaxel combination)
  Plasma PK parameter Vd of POL6326 (balixafortide)
PHASE Ib - PK in terms of apparent half-life (t1/2) | At the end of Cycle 1 (each cycle is 28 days in POL6326 (balixafortide) - eribulin combination and 21 days in POL6326 (balixafortide) - nab paclitaxel combination)
  Plasma PK parameter t1/2 of POL6326 (balixafortide)
PHASE Ib - PK in terms of maximal serum concentration (Cmax) | At the end of Cycle 1 (each cycle is 28 days in POL6326 (balixafortide) - eribulin combination and 21 days in POL6326 (balixafortide) - nab paclitaxel combination)
  Plasma PK parameter Cmax of POL6326 (balixafortide)
PHASE Ib - PK in terms of trough concentrations (Ctrough) | At the end of Cycle 1 (each cycle is 28 days in POL6326 (balixafortide) - eribulin combination and 21 days in POL6326 (balixafortide) - nab paclitaxel combination)
  Plasma PK parameter Ctrough of POL6326 (balixafortide)
PHASE Ib - PK in terms of time of maximum concentration observed (tmax) | At the end of Cycle 1 (each cycle is 28 days in POL6326 (balixafortide) - eribulin combination and 21 days in POL6326 (balixafortide) - nab paclitaxel combination)
  Plasma PK parameter tmax of POL6326 (balixafortide)
PHASE Ib - PK in terms of time to last measurable plasma (tlast) | At the end of Cycle 1 (each cycle is 28 days in POL6326 (balixafortide) - eribulin combination and 21 days in POL6326 (balixafortide) - nab paclitaxel combination)
  Plasma PK parameter tlast of POL6326 (balixafortide)
PHASE 2 - PK in terms of Cmax | At the end of Cycle 1 (each cycle is 28 days in POL6326 (balixafortide) - eribulin combination and 21 days in POL6326 (balixafortide) - nab paclitaxel combination)
  Plasma PK parameter Cmax of POL6326 (balixafortide)
PHASE 2 - PK in terms of Cthrough | At the end of Cycle 1 (each cycle is 28 days in POL6326 (balixafortide) - eribulin combination and 21 days in POL6326 (balixafortide) - nab paclitaxel combination)
  Plasma PK parameter Cthrough of POL6326 (balixafortide)
PHASE 2 - PK in terms of tmax | At the end of Cycle 1 (each cycle is 28 days in POL6326 (balixafortide) - eribulin combination and 21 days in POL6326 (balixafortide) - nab paclitaxel combination)
  Plasma PK parameter tmax of POL6326 (balixafortide)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cortés, MD,PhD, Principal Investigator — International Breast Cancer Center (IBCC), Quiron Group, Barcelona (Spain); Peter Kaufman, MD, Principal Investigator — University of Vermont Medical Center, Burlington (Vermont, USA)